CLINICAL TRIAL: NCT03689946
Title: Effect of Evolocumab on Coronary Artery Plaque Volume and Composition by Coronary CTA (CCTA) and Microcalcification by F18-NaF PET: A Phase 3 Study
Brief Title: Effect of Evolocumab on Coronary Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Daniel S. Berman, Principal Investigator/Chief Nuclear Cardiology and Cardiac Imaging, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54274
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Disease; Hyperlipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias | interventions — evolocumab; Iohexol; Contrast Media; Metoprolol; Adrenergic beta-Antagonists; Nitroglycerin; Vasodilator Agents

STUDY DESIGN:
Intervention Model Description: Early development, single-arm, prospective, open-label study of evolocumab injection in patients with calcified plaque in the coronary artery detected by CCTA. Fifty-five (55) evaluable subjects will be enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Evolocumab, F18-NaF PET, CCTA (Experimental): Evolocumab self-administration for 18 months. Baseline (pre-treatment) and follow-up 18F-NaF PET and CCTA (possible beta-blocker and nitroglycerin, if medically safe).
  Interventions: Drug: Evolocumab; Diagnostic Test: 18F-NaF PET; Diagnostic Test: CCTA; Drug: Omnipaque; Drug: Metoprolol; Drug: Nitroglycerin

INTERVENTIONS:
Drug: Evolocumab — Evolocumab: In patients without homozygous familial hypercholesterolemia (FH), evolocumab will be self-injected as follows: 140mg every 2 weeks or 420mg once a month subcutaneously.
  Patients with homozygous FH will be instructed to administer 420mg subcutaneously once a month by giving 3 injections consecutively within 30 minutes using the single-use prefilled autoinjector.
  Other Names: Repatha®; PCSK9 inhibitor
Diagnostic Test: 18F-NaF PET — 18F-NaF PET: Baseline (pre-treatment) and follow-up dual cardiac and respiratory-gated PET- imaging of the thoracic aorta. Dose of 250 MBq 18F-NaF intravenously.
  Other Names: 18F sodium fluoride; sodium fluoride PET
Diagnostic Test: CCTA — CCTA: Baseline (pre-treatment) and follow-up CCTA. Bolus injection of 80-100 ml contrast (Omnipaque or Visipaque). Possible beta blocker(metoprolol)administered to achieve a target heart ≤70 beats/min (bpm) and/or 0.4 or 0.8 mg of sublingual nitroglycerin administered, if medical safe.
  Other Names: Coronary computed tomography angiography
Drug: Omnipaque — contrast agent for CCTA
  Other Names: contrast
Drug: Metoprolol — beta blocker to optimize heart rate during CCTA
  Other Names: beta blocker
Drug: Nitroglycerin — premedication for CCTA
  Other Names: vasodilator

SUMMARY:
This study will quantify changes in coronary plaque volumes and plaque composition in patients treated with evolocumab.

Previous intravascular ultrasound studies have shown that treatment with a lipid-lowering PCSK9 enzyme inhibitor, such as evolocumab, to be associated with a reduction of the fatty deposits that cause plaque in the arteries, however, it is not known how evolocumab affects specific coronary plaque types and plaque inflammation.

Investigators will use quantitative assessment of non-invasive coronary computed tomography angiography (CCTA) and positron emission tomography (PET)imaging to evaluate functional changes in plaque burden, plaque composition and vascular inflammation before and after treatment with evolocumab.

Investigators propose to show that patients treated with evolocumab in combination with statins demonstrate a greater reduction of coronary non-calcified plaque volume, thereby reducing the number of future cardiac events.

DETAILED DESCRIPTION:
To evaluate the effect of evolocumab, patients who are taking Evolocumab plus another cholesterol-lowering medication (e.g statins), will undergo diagnostic testing including non-invasive coronary CT angiographic (CCTA) scans and positron emission tomography (PET) scans. The CCTA and PET scans will be done before and after being treated with evolocumab.

At the initial visit, standard imaging eligibility screening will take place, as well as blood sampling to test cholesterol levels and presence of proteins (biomarkers) associated with heart disease. A CCTA will be done (if not done for clinical purposes within the past 90 days) and a PET scan with administration of 18F-NaF injection will take place. Patients will receive the first injection of evolocumab and will be taught how to self-inject once or twice a month for 18 months.

After the initial visit, patients will self-inject evolocumab at approximately 6, 12 and 18 months in front of a medical professional for site monitoring and re-training. Labs will be drawn to assess blood components related to heart disease.

Follow-up phone calls will be made at approximately 1,3, 9, 15 months and approximately 3-7 days after their final on-site visit (18 months) to monitor safety and drug adherence.

The final visit (18 months after the initial visit) will involve another PET scan, CCTA and blood collection for biomarker testing.

ELIGIBILITY:
Inclusion Criteria:

* Evidence by CCTA of noncalcified coronary artery plaque (>440 mm3) and thoracic aorta atherosclerosis
* On-label indications for evolocumab treatment which includes the following criteria:

Those who have established cardiovascular disease defined as acute coronary syndrome, history of myocardial infarction, stable angina or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack, or peripheral arterial disease presumed to be of atherosclerotic origin.

Exclusion Criteria:

* Creatinine > 1.5 mg/dL prior to imaging
* History of allergy to iodine contrast agents
* Allergy to evolocumab or any other ingredients contained in study drug
* Pregnancy
* Women who are breastfeeding
* Active atrial fibrillation
* History of coronary artery bypass graft
* Inability to lie flat
* Inability or unwilling to give informed consent
* Major illness or life expectancy <1 year
* Planned coronary revascularization or major non-cardiac surgery in the next 12 months
* Previously or currently on evolocumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Berman, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han D, Tzolos E, Park R, Gransar H, Hyun M, Friedman JD, Hayes SW, Thomson LEJ, Kwan AC, Budoff M, Shah PK, Kwiecinski J, Wetzel S, Findling C, Slomka PJ, Dey D, Tamarappoo BK, Berman DS. Effects of Evolocumab on Coronary Plaque Composition and Microcalcification Activity by Coronary PET and CT Angiography. JACC Cardiovasc Imaging. 2025 May;18(5):589-599. doi: 10.1016/j.jcmg.2025.01.005. Epub 2025 Apr 2. PMID 40178463

RESULTS

PARTICIPANT FLOW:
Groups:
- Evolocumab, F18-NaF PET, CCTA: Evolocumab self-administration for 18 months. Baseline (pre-treatment) and follow-up 18F-NaF PET and CCTA (possible beta-blocker and nitroglycerin, if medically safe).
  Evolocumab: Evolocumab: In patients without homozygous familial hypercholesterolemia (FH), evolocumab will be self-injected as follows: 140mg every 2 weeks or 420mg once a month subcutaneously.
  Patients with homozygous FH will be instructed to administer 420mg subcutaneously once a month by giving 3 injections consecutively within 30 minutes using the single-use prefilled autoinjector.
  18F-NaF PET: 18F-NaF PET: Baseline (pre-treatment) and follow-up dual cardiac and respiratory-gated PET- imaging of the thoracic aorta. Dose of 250 MBq 18F-NaF intravenously.
  CCTA: CCTA: Baseline (pre-treatment) and follow-up CCTA. Bolus injection of 80-100 ml contrast (Omnipaque or Visipaque). Possible beta blocker(metoprolol)administered to achieve a target heart ≤70 beats/min (bpm) and/or 0.4 or 0.8 mg of sublingual nitroglycerin administered, if medical safe.
  Omnipaque: contrast agent for CCTA
  Metoprolol: beta blocker to optimize heart rate during CCTA
  Nitroglycerin: premedication for CCTA
Period: Overall Study
Arm/Group | Evolocumab, F18-NaF PET, CCTA
Started | 55
Completed | 47
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 3
Not completed — Data corruption | 2

BASELINE CHARACTERISTICS:
Population: Of the 55 patients initially enrolled, 3 were lost to follow-up, 3 withdrew consent, and 2 were not included in analysis due to missing imaging information
Arm/Group | Evolocumab, F18-NaF PET, CCTA
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 47
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (4.4)
Risk factors [Count of Participants; unit: Participants]
  Hypertension | 25
  Diabetes | 10
  Hypercholesterolemia | 42
  Current smoker | 1
  Prior CAD history | 4
  Prior CVA history | 1
Medication [Count of Participants; unit: Participants]
  Aspirin | 29
  Statin | 38
  ACEi or ARB | 15
  Beta blocker | 17
  Calcium channel blocker | 7
Plaque volume [Mean (Standard Deviation); unit: mm^3]
  Total plaque volume | 716 (431)
  Non calcified plaque volume | 607 (347)
  Low density non calcified plaque volume | 37 (29)
  Calcified plaque volume | 109 (134)
Cholesterol level [Mean (Standard Deviation); unit: mg/dL]
  Total choleseterol | 155.8 (46.1)
  LDL cholesterol | 82.2 (38.9)
  HDL cholesterol | 47.9 (14.4)
  Triglycerides | 137.6 (81.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Noncalcified Coronary Artery Plaque Volume (NCPV)
Description: Compare NCPV in mm^3 measured on cardiac CT images as analyzed by quantitative software between the two assessments
Time Frame: baseline (pre-treatment) and 18 months after of treatment
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Evolocumab, F18-NaF PET, CCTA
Number analyzed (Participants) | 47
mm^3 | -45 (64)

2. Secondary Outcome: Change in Plaque Composition (Total, Calcified, Low Density Non Calcified)
Description: Chances in volume of type of plaque (total, calcified, low density non calcified) on cardiac CT images as detected by quantitative software between the two assessments
Time Frame: baseline (pre-treatment) and 18 months after of treatment
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Evolocumab, F18-NaF PET, CCTA
Number analyzed (Participants) | 47
mm^3
  Changes in total plaque volume | -5 (97)
  Changes in calcified plaque volume | 40 (56)
  Changes in low density non calcified plaque volume | -17 (24)

ADVERSE EVENTS:
Time Frame: Duration of the study (18 months)
Description: Only adverse events that occurred in at least 5% of the cohort were reported.
Arm/Group | Evolocumab, F18-NaF PET, CCTA
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 3/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evolocumab, F18-NaF PET, CCTA (N=55)
runny nose (Respiratory, thoracic and mediastinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
1. The sample size is small, and the study population was selectively chosen based on baseline plaque burden.
2. Because inclusion criteria focused on plaque burden, the predominantly male population, known to have higher plaque burden, limits the generalizability of the findings.
3. As a single-arm study, the absence of a comparison group receiving statin only treatment or a control group receiving no treatment limits the ability to draw direct comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT03689946/Prot_SAP_000.pdf